CLINICAL TRIAL: NCT01186211
Title: Feasibility of Outpatient Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: OHREB2010262-01H
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis Of Knee
Keywords: knee, joint
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting for elective TKA: Patients will be advised preoperatively about an accelerated path while in hospital that will share many attributes of the standard TOH care map but with several additions, chosen to help reduce pain and hemarthrosis, both felt to be the major impediments to faster recuperation.

SUMMARY:
This proposal outlines the investigators plan to develop, evaluate and implement an accelerated in hospital and community rehabilitation following total knee arthroplasty (TKA) leading to outpatient TKA. The benefits of applying current concepts of improved postoperative analgesia and less invasive surgical technique are expected to improve objective parameters of knee function, increase patients satisfaction, while reducing health care resources requirements as compared with standard rehabilitation. The innovation of combining best practices from orthopaedic sports medicine, Anesthesia, Physiotherapy and Knee reconstruction are expected to realize this goal.

DETAILED DESCRIPTION:
Consecutive patients presenting for elective TKA at the General (Dr. Dervin) will be approached for enrollment.

Dr Dervin will present the study to their patients who are appropriate for the study when first confirmed for joint replacement after clinic assessment. If the patient has indicated that they are interested, the surgeon will inform the research coordinator who will then continue the consenting process. The research coordinator will confirm patient's eligibility to ensure that all inclusion and no exclusion criteria are met. The study will be explained in detail to qualify patients and they will be provided with a copy of the consent form. The consent form will also provide a clause of confidentiality informing patient privacy. All questions will be answered. Patients may also talk to the investigators with any additional questions.

Patients will be advised preoperatively about an accelerated path while in hospital that will share many attributes of the standard TOH care map,but with several additions, chosen to help reduce pain and hemarthrosis, both felt to be the major impediments to faster recuperation.

1. Surgery will be performed with a muscle sparing subvastus approach, chosen because of evidenced decreased pain.
2. Tranexamic acid ( 10 mg/kg) intravenously will be administered to further reduce blood loss at time of tourniquet deflation.
3. The "Game Ready" cold - compression device will be used post operatively to help reduce pain and minimize swelling.

   .

Timeline:

Outcome data collection is expected to be completed by July 1, 2018 to allow for a minimum 6 month follow up.

Outcomes (Metrics):

The outcome measures are provided and are summarized here.

1. Length of stay: We will measure LOS for these patients as compared to a cohort that is comparable in demographics who are being treated concurrently on the service
2. Analgesic use in hospital and at home (where pt will maintain a 28 day pain diary to record analgesics taken and quality of life recovery questions) to be captured with special interest to any opioid sparing effect
3. Physiotherapy will measure the Physical parameters such as range of motion and quadriceps strength during stay and at discharge, 2 weeks , and 1 , 2 and 3 months
4. Patient satisfaction questionnaire outcome: after 6 months to evaluate
5. Health care resource requirement

   1. Physiotherapy visits
   2. Use of mobility aids duration
6. Time to return to work where applicable

Benefits to patient The benefits to the patient will be substantial by improving the pace of recovery with less physical burden and quicker achievement of goals and resumption of normal activity.

ELIGIBILITY:
Inclusion Criteria:

* Must be candidate for Total knee arthroplasty
* Patient of Dr Dervin
* Male or Female
* Age range between 50-75yrs,
* A Subvastus approach can be used

Patients who do not meet any exclusion criteria.

Exclusion Criteria:

* Over 75 of age
* Poor health issues
* Revised surgery on same knee
* Pt with evidence of active infection
* Pt with a BMI larger than 30kg/m2

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The first 20 patients (baseline) will be treated in hospital so we can gauge the potential of inpatient stay and our criteria will be refined. The next group of 20 (intermediate) will be geared toward overnight stay and finally the last 120 patients (full intervention) will be geared for same day discharge using the successful protocol already in place for unicompartment knee arthroplasty (UKA) at TOH.
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2010-11-01 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Pain dairy | 28 days
  measuring pain location,pain intensity, quality of pain, satisfaction with pain management, report any side effects, Quality of recovery, Pain medication schedule, Cryocuff schedule for Game Ready device

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Dervin, MD,MSc,FRCSC, Principal Investigator — OHRI / The Ottawa Hospital
Locations (1):
- The Ottawa General Hospital, Ottawa, Ontario, Canada